CLINICAL TRIAL: NCT01191528
Title: The Comparison of Pulse Oximetry, End-tidal Capnometry, and Integrated Pulmonary Index in Adult Post-operative Patients
Brief Title: The Comparison of Pulse Oximetry, End-tidal Capnometry, and Integrated Pulmonary Index (IPI)
Status: Completed | Type: Observational
Sponsor: Allenmore Hospital (Other)
Responsible Party: Julie Northrup RN, BC, Multicare Health System Allenmore Hospital
Other Study IDs: AH2ESCAP
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Postoperative Care
Keywords: Adult; Post; operative; oximetry; capnometry; Integrated; Pulmonary; Index; End-tidal; Monitoring Respiratory status; post-operative
MeSH Terms: conditions — Erythema Multiforme

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: capnostream 20, Oridian Medical 1987 ltd, Needham MA — Oxygen blood saturation measured by a s sensor that reflects infrared light on oxygenated and deoxygenated arterial blood via a noninvasive, clip on digit sensor connected to a combination capnometer and pulse oximeter monitor.
  End-tidal Carbon dioxide (EtCO2) is measured with a noninvasive nasal cannula sampling line which calculates the EtCO2 from exhaled air. Measurements recorded at 5 second intervals.
  Other Names: OxiMax Nellcor, Covidien, Capnoline, Oridion Medical

SUMMARY:
To compare two ways to test breathing after surgery in acute care setting. One method tests oxygen level of the blood, and one method will test oxygen and the carbon dioxide that is breathed out.

DETAILED DESCRIPTION:
A simple comparison design will be used to compare pulse SpO2 monitoring of respiratory status to a combination of pulse SpO2 monitoring and EtCO2 nasal cannula monitoring with Integrated Pulmonary Index (IPI). Using combination monitor, each subject will serve as their own control with repeated measurements of respiratory rate, SpO2, EtCO2 and IPI at 5 second intervals. Patients will be monitored for a minimum of 8 hours after admission to the acute care unit and through the first night.

Subjects for this study will be a convenience sample post-operative in-patients admitted to 2 East after surgery at Allenmore Hospital/Multicare Health System a 75 bed community facility.

ELIGIBILITY:
Inclusion criteria:

* Age greater than 18
* Increased Body Mass Index (BMI) > 31
* History of chronic obstructive pulmonary disease (COPD)
* History of Sleep Apnea

Exclusion criteria:

* Respiratory failure
* Isolation requirements
* Surgical patients admitted to 2 West or ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample post-operative in-patients admitted to 2 East at Allenmore Hospital/multicare Health system a 75 bed community facility.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Northrup, ADN, BC, Principal Investigator — Multicare Health System-Allenmore Hospital; Jennifer Spotted-Horse, MS,BSN,OCN, Principal Investigator — Multicare Health System-Allenmore Hospital; Dawn Fox, RN, Principal Investigator — Multicare Health System-Allenmore Hosptial; David Lechich, RN, Principal Investigator — Multicare Health System-Allenmore Hospital; Joan Fortune, RN, Principal Investigator — Multicare Health System Allenmore Hospital; Katy Rogers, RN, Principal Investigator — Multicare Health System, Allenmore Hospital; Lynn Arnold, RN, Principal Investigator — Multicare Health System Allenmore Hospital; Lisa Ettlin-Porter, BSN,RN,CCRN, Principal Investigator — Multicare Health System Allenmore Hospital; Dee Harris, BS,RRT,RPFT, Principal Investigator — Multicare Health System Allenmore Hospital; Colleen Doherty, PhD(c),RN, Principal Investigator — Consultant-Multicare Health System Allenmore Hospital
Locations (1):
- Allenmore Hospital, Tacoma, Washington, United States